CLINICAL TRIAL: NCT02328976
Title: Hypothalamus Connectivity in Chronic and Episodic Migraine in Headache-free Period: A Resting State Functional Magnetic Resonance Imaging Study
Brief Title: Hypothalamus Connectivity in Chronic and Episodic Migraine
Acronym: HYPOTHAMIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13 197 02
Record Dates: First submitted 2014-02-25; First posted 2014-12-31 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chronic migraineurs (Experimental): functional Magnetic Resonance Imaging (fMRI) analysis to compare connectivity of hypothalamus
  Interventions: Other: functional Magnetic Resonance Imaging (fMRI)
- Episodic migraineurs (Experimental): functional Magnetic Resonance Imaging (fMRI) analysis to compare connectivity of hypothalamus
  Interventions: Other: functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Other: functional Magnetic Resonance Imaging (fMRI) — both chronic and episodic patients with migraine have a specific functional Magnetic Resonance Imaging (fMRI)

SUMMARY:
The purpose is to compare, using functional magnetic resonance imagery in resting-state, the connectivity of the hypothalamus in 2 groups of migraineurs. The first group is composed of chronic migraineurs, studied outside a migraine attack and is compared to gender- and age- matched episodic migraineurs with very few attacks per month and studied in the attack-free period. The primary outcome will be the connectivity index of the hypothalamus to brainstem areas activated during migraine attacks and to the trigeminal-cervical complex.

DETAILED DESCRIPTION:
Functional magnetic resonance imagery allows identification of correlations during rest between remote brain areas (functional connectivity) through their highly correlated low-frequency spontaneous fluctuations. This technique is interesting because it is atraumatic, takes place in resting condition, without administration of substances. Only one study of connectivity with functional magnetic resonance imagery in resting state, in headache-free period of migraine, has shown differences in the connection of the periaqueductal gray matter to the pain matrix in migraineurs and controls. Our region of interest is the hypothalamus because our group demonstrated activation in this area during migraine attacks and we hypothesised that the hypothalamus could trigger migraine attacks. We want to compare 2 groups of migraineurs. The first group is composed of chronic migraineurs with >15 days with headache per month, compared to the 2nd group composed of age- and gender-matched episodic migraineurs with < 4 days of migraine per month, without prophylactic treatment. Our purpose is to study the connectivity of the hypothalamus to midbrain and pons areas activated in previous studies using positon emission tomography (PET) in spontaneous migraine attacks. The connectivity of the hypothalamus with the trigeminal-cervical complex, conveying the pain from cranial vasculature and dura-mater playing a major role in migraine attack, has never been studied before, mainly for anatomical reasons. Our secondary purpose is to study the connectivity of the hypothalamus with the pain matrix and the possible correlations with depression, allodynia and attack treatment overuse.

The primary outcome is the connectivity index of the hypothalamus to the midbrain and pons area known to be activated in migraine attacks and the trigeminal-cervical complex The secondary outcome is the connectivity index of the hypothalamus with the pain matrix (thalamus, sensitive-motor cortex, cingular cortex) This study is a comparative monocentric pathophysiological study of patients with migraine.

ELIGIBILITY:
Inclusion criteria:

* patients fulfilling international criteria of chronic migraine (with or without medication overuse)
* age 18-65 years,
* with or without migraine prophylactic treatment (unchanged for 3 months). Inclusion criteria of patients with episodic migraine are: age- and- gender matched patients, fulfilling international criteria: migraine without aura, with 4 days with migraine/month, without prophylactic treatment, without history of chronic migraine

Exclusion criteria:

* evolutive severe coexistent chronic disease,
* MRI contra-indications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
connectivity index measure | 3 months
  connectivity between hypothalamus and nociception areas

CONTACTS AND LOCATIONS:
Overall Officials: Nelly FABRE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denuelle M, Fabre N. Functional neuroimaging of migraine. Rev Neurol (Paris). 2013 May;169(5):380-9. doi: 10.1016/j.neurol.2013.02.002. Epub 2013 Apr 18. PMID 23602115
- [Result] Lerebours F, Boulanouar K, Barege M, Denuelle M, Bonneville F, Payoux P, Larrue V, Fabre N. Functional connectivity of hypothalamus in chronic migraine with medication overuse. Cephalalgia. 2019 Jun;39(7):892-899. doi: 10.1177/0333102419833087. Epub 2019 Mar 5. PMID 30836766